CLINICAL TRIAL: NCT04271722
Title: Clinical Evaluation of Cervical Ripening in the Outpatient Setting Using Mifepristone Versus Balloon Catheter: a Randomized Controlled Trial
Brief Title: Clinical Evaluation of Cervical Ripening in the Outpatient Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Hospitalar Lisboa Norte (Other)
Responsible Party: Principal Investigator, Maria de Carvalho Afonso, Medical Doctor, Phd Student, Centro Hospitalar Lisboa Norte
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020OBST1
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Labor; Forced or Induced, Affecting Fetus or Newborn; Labor Onset and Length Abnormalities
Keywords: cervical ripening; mifepristone; balloon catheter
MeSH Terms: interventions — Cervical Ripening

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mifepristone (Experimental): Mifepristone 200mg 24hours before the induction day
  Interventions: Other: Cervical ripening
- Balloon catheter (Active Comparator): Balloon catheter with 40ml placed 24hours before the induction day
  Interventions: Other: Cervical ripening

INTERVENTIONS:
Other: Cervical ripening — Subjects will undergo cervical ripening in the outpatient setting. The patients will then be scheduled to return the next morning for induction of labor.

SUMMARY:
A randomized controlled trial of mifepristone 200mg vs balloon catheter for cervical ripening.

DETAILED DESCRIPTION:
Artificial induction of labour is currently required in 25-30% of all pregnancies, in high-resource countries. While the pharmacological modifications to the collagen matrix of the cervix, that allow it to dilate (cervical ripening) occur spontaneously in many women, allowing labour to be induced with oxytocin, in others the process needs to be triggered artificially. Cervical ripening is traditionally accomplished with prostaglandins or mechanical agents, in processes that typically require 12-24 hours of hospital stay. More recently, a limited number of hospitals have shifted towards starting the process in house, but then allowing women to return home and be re-evaluated on the following day.

The main aims this study is to compare efficacy and patient satisfaction of mifepristone vs balloon catheter for cervical ripening.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman scheduled for induction of labor.
* Age between 18 and 45 years.
* Understanding and capable to sign informed consent.
* Singleton pregnancy.
* Gestational age ≥ 37 0/7 weeks.
* Live fetus in cephalic presentation.
* Intact membranes
* Bishop score < 6
* Estimated fetal weight < 4500g
* Without contraindication to vaginal delivery
* No major fetal anomaly

Exclusion Criteria:

* Previous cesarean section or myomectomy
* Hypertension
* Diabetes
* Thyroid disease
* Maternal conditions with high risk of placental insufficiency

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Bishop score ≥6 or spontaneous labour | 24 hours
  Proportion of patients (%) with Bishop score ≥6 or spontaneous labour 24 hours after intervention

SECONDARY OUTCOMES:
Mean of gain in Bishop score | 24 hours
  Mean of gain in Bishop score from intervention to hospital admission
Time frame between intervention and active phase of labour | 1-2 days
  Time frame between intervention and active phase of labour (min)
Time of Vaginal Delivery | 2-4days
  Delivery time frame in mins from intervention
Number of Participants with vaginal delivery within 24hrs | 1-2days
  Rate of vaginal deliveries within 24 hours since admission to hospital (%)
Vaginal delivery within 48hrs | 1-2days
  Rate of vaginal deliveries within 48 hours since admission to hospital (%)
Pharmacological agents for labor induction (Prostaglandins, Oxytocin) | 1-2days
  Rate of women that required pharmacological cervical ripening agents (%) requirement (%)
Operative deliveries | 1-4days
  Proportion of patients that delivered vaginal by forceps assistance or vacuum (%) assistance.
Cesarean deliveries | 1-4days
  Proportion of patients that delivered by cesarean (%).
Analgesia requirement | 24 hours
  Rate of women who require any analgesia during cervical ripening process (%)
Vaginal bleeding | 24 hours
  Rate of women who had vaginal bleeding during cervical ripening process (%)
Reduced fetal movements | 24 hours
  Rate of women who had reduced fetal movements during cervical ripening process (%)
Non reassuring fetal status | 24 hours
  Rate of women who had non reassuring fetal status(CTG) during cervical ripening process (%)
Patient Satisfaction: questionnaire | 1-4days
  Patient satisfaction associated with intervention used for cervical ripening from patient questionnaire

OTHER OUTCOMES:
Neonatal Intensive Care Unit admission | 1-30 days
  Rate of newborns admitted in Neonatal Intensive Care Unit (%)
Postpartum haemorrhage | 1-7 days
  Rate of women with postpartum haemorrhage (%)
5 minute apgar score <7 | 1-4 days
  Rate of newborns with 5 minute apgar score <7 (%)
Metabolic acidosis(pH< 7.00 e BD > 12 mmol/l) | 1-4 days
  Rate of metabolic acidosis (pH< 7.00 e BD > 12 mmol/l) (%)
Neonatal mortality | 1-7days
  Rate of neonatal mortality (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar Lisboa Norte, Lisbon, Portugal

REFERENCES:
- [Background] Diederen M, Gommers J, Wilkinson C, Turnbull D, Mol B. Safety of the balloon catheter for cervical ripening in outpatient care: complications during the period from insertion to expulsion of a balloon catheter in the process of labour induction: a systematic review. BJOG. 2018 Aug;125(9):1086-1095. doi: 10.1111/1471-0528.15047. Epub 2018 Jan 10. PMID 29211328
- [Background] Heikinheimo O, Kekkonen R, Lahteenmaki P. The pharmacokinetics of mifepristone in humans reveal insights into differential mechanisms of antiprogestin action. Contraception. 2003 Dec;68(6):421-6. doi: 10.1016/s0010-7824(03)00077-5. PMID 14698071
- [Background] Smith R, Smith JI, Shen X, Engel PJ, Bowman ME, McGrath SA, Bisits AM, McElduff P, Giles WB, Smith DW. Patterns of plasma corticotropin-releasing hormone, progesterone, estradiol, and estriol change and the onset of human labor. J Clin Endocrinol Metab. 2009 Jun;94(6):2066-74. doi: 10.1210/jc.2008-2257. Epub 2009 Mar 3. PMID 19258402
- [Background] Ceccaldi PF, Saada J, Nicolas M, Ducarme G, Blot P, Guibourdenche J, Luton D. Modulation of free corticotrophin-releasing hormone, adrenal and placental steroid hormone levels induced by mifepristone during pregnancy. Fetal Diagn Ther. 2012;32(4):267-70. doi: 10.1159/000338927. Epub 2012 Jul 4. PMID 22759411
- [Background] Rodger MW, Baird DT. Pretreatment with mifepristone (RU 486) reduces interval between prostaglandin administration and expulsion in second trimester abortion. Br J Obstet Gynaecol. 1990 Jan;97(1):41-5. doi: 10.1111/j.1471-0528.1990.tb01714.x. PMID 2407284
- [Background] Urquhart DR, Bahzad C, Templeton AA. Efficacy of the antiprogestin mifepristone (RU 486) prior to prostaglandin termination of pregnancy. Hum Reprod. 1989 Feb;4(2):202-3. doi: 10.1093/oxfordjournals.humrep.a136872. PMID 2918074
- [Background] Elliott CL, Brennand JE, Calder AA. The effects of mifepristone on cervical ripening and labor induction in primigravidae. Obstet Gynecol. 1998 Nov;92(5):804-9. doi: 10.1016/s0029-7844(98)00284-1. PMID 9794673
- [Background] Yelikar K, Deshpande S, Deshpande R, Lone D. Safety and Efficacy of Oral Mifepristone in Pre-induction Cervical Ripening and Induction of Labour in Prolonged Pregnancy. J Obstet Gynaecol India. 2015 Jul;65(4):221-5. doi: 10.1007/s13224-014-0584-6. Epub 2014 Jul 11. PMID 26243986
- [Background] Baev OR, Rumyantseva VP, Tysyachnyu OV, Kozlova OA, Sukhikh GT. Outcomes of mifepristone usage for cervical ripening and induction of labour in full-term pregnancy. Randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2017 Oct;217:144-149. doi: 10.1016/j.ejogrb.2017.08.038. Epub 2017 Sep 1. PMID 28898687
- [Background] Vogel JP, Osoti AO, Kelly AJ, Livio S, Norman JE, Alfirevic Z. Pharmacological and mechanical interventions for labour induction in outpatient settings. Cochrane Database Syst Rev. 2017 Sep 13;9(9):CD007701. doi: 10.1002/14651858.CD007701.pub3. PMID 28901007